CLINICAL TRIAL: NCT04152629
Title: A Phase IV, Real World, Open-label, Multi-centre Study on the Use of FOQUEST® (Methylphenidate Hydrochloride Controlled-release Capsules) for the Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in Pediatric and Adult Patients
Brief Title: Real World Evidence of the Efficacy and Safety of FOQUEST
Acronym: reFOQus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Purdue Pharma, Canada (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN-MA-FOQ-001
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit-Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- FOQUEST adults (Experimental): adult (≥18 years or older) patients with ADHD receiving FOQUEST (controlled-release methylphenidate 25 mg, 35 mg, 45 mg, 55 mg, 70 mg, 85 mg, or 100 mg/day)
  Interventions: Drug: Methylphenidate Hydrochloride
- VYVANSE adults (Active Comparator): adult (≥18 years or older) patients with ADHD receiving VYVANSE (lisdexamfetamine 10 mg, 20 mg, 30 mg, 40 mg, 50 mg or 60 mg/day)
  Interventions: Drug: Lisdexamfetamine Dimesylate
- FOQUEST pediatric (Experimental): pediatric (6 to 17 years old) patients with ADHD receiving FOQUEST (controlled-release methylphenidate 25 mg, 35 mg, 45 mg, 55 mg or 70 mg/day)
  Interventions: Drug: Methylphenidate Hydrochloride
- VYVANSE pediatric (Active Comparator): pediatric (6 to 17 years old) patients with ADHD receiving VYVANSE (lisdexamfetamine 10 mg, 20 mg, 30 mg, 40 mg, 50 mg or 60 mg/day)
  Interventions: Drug: Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride — CR Methylphenidate Hydrochloride given once daily (25 mg, 35 mg, 45 mg, 55 mg, 70 mg, 85 mg or 100 mg)
  Other Names: FOQUEST; ADHANSIA XR
  Arms: FOQUEST adults; FOQUEST pediatric
Drug: Lisdexamfetamine Dimesylate — Lisdexamfetamine Dimesylate given once daily (10 mg, 20 mg, 30 mg, 40 mg, 50 mg or 60 mg)
  Other Names: VYVANSE
  Arms: VYVANSE adults; VYVANSE pediatric

SUMMARY:
This study is a four-month, phase IV, open-label study of ADHD symptomatology and functional outcomes in pediatric (6 to 17 years old) and adult (≥18 years or older) patients with ADHD treated with FOQUEST or VYVANSE.

DETAILED DESCRIPTION:
After giving written, informed consent or assent (for patients <18 years old), patients will be screened to ascertain their suitability for the study according to the patient selection criteria (Section 4). Based on clinician assessment, patients will be assigned to receive either FOQUEST or VYVANSE. Patients will be titrated to their optimal dose of ADHD medication based on Investigator judgement. At monthly visits, patients will have their ADHD symptomatology evaluated by the Investigator (ADHD-Rating Scale-DSM 5 Version [ADHD-RS-5]) and will complete questionnaires on functional outcomes (Weiss Functional Impairment Ratings Scale - Parent [WFIRS-P] or Weiss Functional Impairment Ratings Scale - Self [WFIRS-Self]), morning and evening behaviours (Daily Parent Rating of Evening and Morning Behaviours - Revised [DPREMB-R] or Adult ADHD Quality of Life Rating Scale - Revised [AAQoL-R]) and Patient Sleep & Satisfaction survey (PSS). Safety will be evaluated through non-directed spontaneous adverse event (AE) reporting. Patients will be monitored for signs of suicide-related behavior, as per standard of care. A post-study safety follow-up phone call (conducted between 7 and 14 days post-last visit) will assess patients for any adverse events that occur following their last dose of medication received as part of the study. Following the last dose of study medication, the patient's continuing, post-study ADHD treatment will be based on Investigator discretion and standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric: Male or non-pregnant, non-nursing female patients the age of 6 to less than 18. Adults: Male or non-pregnant, non-nursing female patients the age of 18 or older.
2. Diagnosed with ADHD (inattentive, hyperactive or combined-type) who are deemed eligible to receive treatment with FOQUEST or VYVANSE, as per the respective Product Monograph.
3. Mentally and physically competent to provide informed consent, or assent and able and willing to comply with the study protocol, including the study duration.

Exclusion Criteria:

Potential patients who meet any of the contraindications or warnings detailed in the respective Canadian Product Monographs are excluded from participation in the study:

1. Having a true allergy to methylphenidate or amphetamines or sympathomimetic amines, history of serious adverse reactions to methylphenidate or amphetamines or be known to be non-responsive to methylphenidate or amphetamine treatment. Non-response is defined as methylphenidate or amphetamine use at various doses for a phase of at least four weeks at each dose with little or no clinical benefit in the past 10 years.
2. Females of child-bearing potential (FOCP) who are pregnant, planning on becoming pregnant or breast feeding.
3. Having a history of hyperthyroidism, thyrotoxicosis, advanced arteriosclerosis, severe renal insufficiency or glaucoma.
4. Having structural cardiac abnormalities, symptomatic cardiovascular disease or moderate to severe hypertension.
5. Currently, or within the past 14 days, receiving MAO inhibitors.
6. Having a primary diagnosis of bipolar disorder, as assessed at Visit 1.
7. Currently receiving any investigational drug, or have received an investigational drug in the previous month.
8. Having a history of drug or alcohol abuse or dependence.
9. Currently considered a suicide risk by the Investigator.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Change in ADHD Rating Scale Total Score | Change from Baseline ADHD Rating Scale Total Score at 4 months
  The ADHD Rating Scale DSM-5 (ADHD-RS-5) is a clinician-rated scale that reflects current symptoms of ADHD based on DSM-5 criteria. It is a global assessment that measures the severity of symptoms from visit to visit, but is not utilized to assess symptoms of ADHD over the course of the day. The ADHD-RS-5 consists of 18 items that are grouped into two subscales (hyperactivity/impulsivity, and inattention). Higher score means higher frequency and severity of symptoms.

SECONDARY OUTCOMES:
Non-Inferiority Comparison between Treatments in Change in ADHD Rating Scale Total Score | Change from Baseline ADHD Rating Scale Total Score at 4 Months
  The ADHD Rating Scale DSM-5 (ADHD-RS-5) is a clinician-rated scale that reflects current symptoms of ADHD based on DSM-5 criteria. It is a global assessment that measures the severity of symptoms from visit to visit, but is not utilized to assess symptoms of ADHD over the course of the day. The ADHD-RS-5 consists of 18 items that are grouped into two subscales (hyperactivity/impulsivity, and inattention). Higher score means higher frequency and severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (11):
  - Matheson Centre for Mental Health Research & Education, University of Calgary, Calgary, Alberta
  - Adult ADHD Centeres at Pacific Coast Recovery Care, Burnaby, British Columbia
  - Medical Arts Health Research Group, Burnaby, British Columbia
  - The Kids Clinic Inc., Ajax, Ontario
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Pediatric Institute of Excellence, Etobicoke, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Center for Pediatric Excellence, Ottawa, Ontario
  - ADDClinic Windsor, Windsor, Ontario
  - Recherche Clinique Sigma Inc, Québec, Quebec
  - Alpha recherche clinique, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No